CLINICAL TRIAL: NCT00202930
Title: Use of Rituximab in Opsoclonus-Myoclonus in Children With Neuroblastoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed early due to low accrual.
Sponsor: Jean M. Tersak, M.D. (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Jean M. Tersak, M.D., Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB0405652
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Neuroblastoma; Opsoclonus-myoclonus
Keywords: neuroblastoma; Opsoclonus-myoclonus; rituximab
MeSH Terms: conditions — Neuroblastoma; Opsoclonus-Myoclonus Syndrome | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rituximab (Other): Single Arm
  Interventions: Drug: anti-CD20 (Rituximab)

INTERVENTIONS:
Drug: anti-CD20 (Rituximab) — 4 weekly doses of IV rituxan at 375 mg/m2 on days 1, 8, 15 and 22
  Other Names: Rituxan

SUMMARY:
The purpose of this study is to evaluate the feasibility of giving four weekly doses of Rituximab (anti-CD20 antibody) in the treatment of children with refractory neuroblastoma associated opsoclonus-myoclonus. Patients must have continued symptoms of opsoclonus, myoclonus and or ataxia despite surgical resection and a minimum of one month of steroid therapy. Evaluations include clinical symptoms of opsoclonus-myoclonus and ataxia as well as detailed evaluation of learning and development.

DETAILED DESCRIPTION:
Opsoclonus-myoclonus ataxia syndrome (OMS) is a rare immune mediated paraneoplastic syndrome that occurs in approximately 2 to 3% of children with neuroblastoma. Children with neuroblastoma associated opsoclonus-myoclonus tend to have a favorable prognosis from the standpoint of the cure of their cancer. Unfortunately,approximately two-thirds of this subgroup of patients are left with long term sequellae of the syndrome, including residual symptoms of opsoclonus, myoclonus, ataxia, learning difficulties and disturbance of sleep and mood.

Multiple lines of evidence indicate an immune mechanism to this rare disorder. This includes occurence of OMS in the post-infectious state, aggressive lymphocytic infiltration of the tumor in children with OMS, and documented responses to therapries that act through suppression of the immune system.

The current study utilizes four weekly doses of anti-CD 20 antibody (rituximab) to treat children with refractory OMS. Refractory disease is defined as continued symptoms of OMS despite surgical resection of the tumor and a minimum of one month of steroid therapy.

All patients have baseline OMS evaluation and detailed neurocognitive testing with all studies being repeated at the completion of the four weekly infusions. OMS testing is repeated at Month 3. OMS testing and detailed neurocognitive testing is conducted at 6 months intervals until 2 years from the initial infusion.

The goal of the study is to utilize this novel therapy to improve long term neurologic and neurodevelopmental outcome in children with refratory neuroblastoma associated opsoclonus-myoclonus.

ELIGIBILITY:
Inclusion Criteria:

Pathologic confirmation of diagnosis of neuroblastoma Surgical resection of primary tumor Symptoms of OMS despite a minimum of one month of steroid therapy Must meet all laboratory criteria to demonstrate adequate organ function -

Exclusion Criteria:

Patients currently receiving systemic chemotherapy for treatment of neuroblastoma Patients with documented active infection Patients who are HIV, Hep B or Hep C positive Organ toxicity from any prior therapy or surgical intervention must be resolved prior to study entry

-

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2005-07; Primary Completion 2008-12 (Actual); Study Completion 2009-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean M Tersak, M.D., Principal Investigator — Children's Hospital of Pittsburgh Department of Hematology Oncology and BMT

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab: Participants received 4 weekly doses of IV rituxan at 375 mg/m^2 on days 1, 8, 15 and 22
Period: Overall Study
Arm/Group | Rituximab
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 4
OMS Evaluation Scale of Motor-Performance. [Mean (Full Range); unit: units on a scale] — OMS Evaluation Scale of Motor-Performance. This scoring system utilizes a scale of 0 to 3, with 0 being unaffected by OMS, and 3 representing those with severe impairment. OMS testing will be scored by two independent scorers who have special expertise in the evaluation and management of children with neurologic disorders. The mean of these scores will be obtained, and a standard error of the mean reported.
  units on a scale | NA [NA to NA] — The raw data for OMS scoring is at the NIH in the offices of Dr. Nina Schor, MD PhD. She was the responsible neurology investigator in this study. The trial closed early due to low accrual and did not enroll adequate numbers to conduct detailed statistical analysis of the raw data. Due to the pandemic and discontinuation of in person activities, a decision was made by the NIH to undertake extensive renovations of the facility. Dr. Schor is unable to access them due to construction.

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Using 4 Weekly Rituximab Infusions
Description: To evaluate the feasibility of using 4 weekly Rituximab infusions in the treatment of children with neuroblastoma associated opsoclonus-myoclonus syndrome (OMS). The first infusion involved a slow up titration from an initial rate of 0.5 mg/kg/hour to a maximum of 400 mg/hour. If well tolerated, the subsequent infusions were administered at a starting rate of 1 mg/kg/hour to a maximum of 100 mg/hour for the first hour. In the absence of adverse reaction doses were escalated by 1 mg/kg/hour (maximum 100 mg increase per hour) every 30 minutes to a maximum rate of 400 mg/hour. If hypersensitivity or infusion related events occurred, the infusion was temporarily interrupted and resumed at 50% of the previous rate if reaction resolves. The number of participants for whom the study dosing was feasible is reported.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab
Number analyzed (Participants) | 4
Participants | 4

2. Primary Outcome: Toxicity of Rituximab
Description: The trial was to be terminated early for any grade 3 or 4 toxicity that did not resolve in 2 of the first 5 patients treated, or for any infusion related death. The number of participants who experienced these events [grade 3 or 4 toxicity that did not resolve in 2 of the first 5 patients treated, or for any infusion related death] is reported.
Time Frame: Individuals were followed for adverse events until day 270
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab
Number analyzed (Participants) | 4
Participants | 0

3. Secondary Outcome: OMS Evaluation Scale of Motor-Performance
Description: OMS Evaluation Scale of Motor-Performance This scoring system utilizes a scale of 0 to 3, with 0 being unaffected by OMS, and 3 representing those with severe impairment. OMS testing will be scored by two independent scorers who have special expertise in the evaluation and management of children with neurologic disorders. The mean of these scores will be obtained, and a standard error of the mean reported.
Time Frame: Baseline, following the four infusions, at months 3, 6, 12, 18 and 24 following the first infusion.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Rituximab
Number analyzed (Participants) | 4
score on a scale | NA [NA to NA] — The raw data for OMS scoring is at the NIH in the offices of Dr. Nina Schor, MD PhD. She was the responsible neurology investigator in this study. The trial closed early due to low accrual and did not enroll adequate numbers to conduct detailed statistical analysis of the raw data. Due to the pandemic and discontinuation of in person activities, a decision was made by the NIH to undertake extensive renovations of the facility. Dr. Schor is unable to access them due to construction.

4. Secondary Outcome: Human-anti-chimeric Antibody (HACA) Development
Description: Blood samples to be evaluated for the occurrence of antibody formation and potential effect on pharmacokinetic profiles.
Time Frame: Baseline; 3, 6, 9 months post treatment
Population: These studies were unable to be performed due to withdraw of funding from the study sponsor. 0 of 4 patients participated.
Arm/Group | Rituximab
Number analyzed (Participants) | 0

5. Secondary Outcome: Peripheral B Cell Depletion
Description: B cell depletion was measured through analysis of serum IgG levels. The number of participants who experienced B cell depletion is reported.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab
Number analyzed (Participants) | 4
Participants | 0

ADVERSE EVENTS:
Time Frame: In addition to outlined in-office evaluations, telephone contact to inquire regarding hospitalizations and adverse event questioning will be performed at days 60, 120 and 270 due to the length of time between scheduled testing.
Arm/Group | Rituximab
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (N=4)
Febrile illness with upper respiratory symptoms and dehydration (General disorders) | 1 (1) — Patient was admitted for community acquired febrile illness with upper respiratory symptoms and dehydration. Blood cultures were negative. Patient recovered and was discharged to home two days following admission. Event was unrelated to study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No